CLINICAL TRIAL: NCT03280160
Title: A Multicenter, Non-randomized, Open Label Study to Evaluate the Efficacy and Security of Ibrutinib Followed by Ibrutinib Consolidation in Combination With Ofatumumab in Previously Untreated Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Protocol GELLC-7: Ibrutinib Followed by Ibrutinib Consolidation in Combination With Ofatumumab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELLC-7
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Ibrutinib 140 MG Oral Capsule [Imbruvica] — Ibrutinib will be administered orally 420 mg (3 x 140 mg capsules) once daily on a continuous schedule on an outpatient basis until disease progression or unacceptable toxicity.
  After 12 cycles of ibrutinib, patients that do not achieve a complete response (CR) will be treated with the combination of ibrutinib and ofatumumab. Patients in CR after 12 cycles of ibrutinib will continue with ibrutinib alone.
  Ofatumumab will be administered by IV infusion, 300mg on Day 1 and 1,000 mg on Day 8 of cycle 13, followed by 5 monthly infusions of 1,000 mg (Day 1 of subsequent 28-day cycles for cycles C14, C15, C16, C17, and C18).
  A treatment cycle will be defined as lasting 28 days
  Other Names: Ofatumumab

SUMMARY:
Based on the promising results obtained with ibrutinib as single agent, the results obtained with ibrutinib in combination with ofatumumab in a previous phase I/IIb study (Jaglowski 2015), and since data from in vitro studies do not support a synergistic effect of the combination of ibrutinib and anti-CD20 mAbs, we propose a chemotherapy-free combined strategy based on ibrutinib monotherapy as front line treatment for patients with CLL, with the addition of a consolidation phase with ofatumumab in patients not attaining CR under ibrutinib in order to improve the quality of their response. Since median time to CR with ibrutinib was nearly 12 months, patients will be evaluated at this time point, and those patients not in CR will add consolidated treatment with Ofatumumab. Thus, this multi-center, non-randomized phase 2 study is designed to evaluate the efficacy and safety of ibrutinib alone or in combination with Ofatumumab in patients no attaining CR under ibrutinib as front-line therapy for patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Multicenter, non- randomized, open-label, double agent, phase II study of the Spanish Group of CLL (GELLC).

Patients with untreated CLL/SLL. Ibrutinib will be administered orally 420 mg (3 x 140 mg capsules) once daily on a continuous schedule on an outpatient basis until disease progression or unacceptable toxicity.

After 12 cycles of ibrutinib, patients that do not achieve a complete response (CR) will be treated with the combination of ibrutinib and ofatumumab. Patients in CR after 12 cycles of ibrutinib will continue with ibrutinib alone.

Ofatumumab will be administered by IV infusion, 300mg on Day 1 and 1,000 mg on Day 8 of cycle 13, followed by 5 monthly infusions of 1,000 mg (Day 1 of subsequent 28-day cycles for cycles C14, C15, C16, C17, and C18).

A treatment cycle will be defined as lasting 28 days. Patients will be treated with ibrutinib, within the study frame, until progression, unacceptable toxicity or cycle C42 of treatment).

All patients still on study treatment at the time of cycle C42, or if the study is stopped early, will be transitioned to prescribed ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with previously untreated CLL or SLL defined following IWCLL criteria (Hallek, 2008).
* Must understand and voluntarily sign an informed consent form.
* Age ≥ 18 years at the time of signing the informed consent form and must be able to adhere to the study visit schedule and other protocol requirements.
* Must have a documented diagnosis of CLL or SLL [IWCLL guidelines for diagnosis and treatment of CLL (Hallek, 2008)] meeting at least one of the following criteria:

Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.

Massive (i.e. > 6 cm below the left costal margin) or progressive or symptomatic splenomegaly.

Massive nodes (i.e. > 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.

Progressive lymphocytosis with an increase of > 50% over a 2-month period, or lymphocyte doubling time (LDT) of less than 6 months.

A minimum of any one of the following disease-related symptoms: unintentional weight loss ≥ 10% within the previous 6 months, significant fatigue (i.e., ECOG PS 2; cannot work or unable to perform usual activities), fevers of greater than 38.0° C or 100.5F for 2 or more weeks without other evidence of infection, or night sweats for more than 1 month without evidence of infection

* Physically fit patients defined as CIRS < 6 (CIRS Scale, Appendix E).
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.
* All sexually active subjects with the capacity to reproduce (male and female) must use high-efficacy contraceptive methods during the course of the study. These restrictions apply for 12 months after the last dose of ofatumumab or 3 months after the last dose of ibrutinib, whichever happens later. High-efficacy contraceptive methods include:

Total abstinence when consistent with the subject's typical and preferred lifestyle (periodic abstinence [e.g. calendar methods, ovulation, symptothermal and post-ovulation methods] and the withdrawal method are not acceptable contraceptive methods).

Female sterilisation defined as surgical hysterectomy, bilateral oophorectomy, or tubal ligation at least six weeks prior to the study treatment (a simple oophorectomy does not meet the definition of female sterilisation).

Male sterilisation (at least six months before screening). A man who has undergone a vasectomy must be the only partner who is a study subject.

Combination of two of the following methods (a+b or a+c or b+c):

1. Use of oral, injected or implanted hormonal contraceptives, or other hormonal contraceptive methods that have a comparable efficacy (failure rate < 1%), for example, hormonal vaginal ring or transdermal hormonal contraceptive. If an oral contraceptive is used, women must use the same pill for a minimum of three months before taking the study treatment.
2. Placement of an intrauterine device (IUD) or an intrauterine system (IUS).
3. Barrier contraceptive methods: condom or cervical cap (cervical/vault diaphragm or cap) with foam/gel/film/spermicidal cream/vaginal suppository.

   * Female subjects of childbearing potential must have a negative pregnancy test at screening. Females of child bearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression

Exclusion Criteria:

* Prior treatment for CLL or SLL.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form.
* Systemic infection that has not resolved prior to initiating study treatment in spite of adequate anti-infective therapy.
* Pregnant or lactating females.
* Participation in any clinical study or having taken any investigational therapy within 28 days prior to initiating study therapy.
* Central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging.
* Prior history of malignancies, other than CLL, unless the patient has been free of the disease for ≥ 3 years.

Exceptions include the following:

Basal cell carcinoma of the skin Squamous cell carcinoma of the skin Carcinoma in situ of the cervix Carcinoma in situ of the breast Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)

* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection.
* Any of the following laboratory abnormalities:

Serum creatinine ≥ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft-GaultAppendix C) ≤ 40 mL/min/1.73m2 Absolute neutrophil count (ANC) < 1.0 X 109/L, unless secondary to bone marrow involvement by CLL.

Platelet count <100,000/mm3 or <50,000/mm3 if bone marrow involvement independent of transfusion support in either situation Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetictransaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) >3 x upper limit of normal (ULN).

Serum total bilirubin > 1.5 x ULN, except in cases of Gilbert's syndrome.

* Presence of autoimmune haemolytic anemia or autoimmune thrombocytopenia.
* Disease transformation [i.e. Richter's Syndrome (lymphomas) or prolymphocytic leukemia.
* Major surgery within the last 28 days prior to registration.
* History of stroke or intracranial hemorrhage within 6 months prior to enrolment.
* Currently active, clinically significant cardiovascular disease or a history of myocardial infarction within 3 months prior to enrolment.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists within 28 days of first dose of study drug.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of response rate | 18 months
  To determine the complete response rate obtained with the combination of Ibrutinib and ofatumumab

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital Son Espases (Son Dureta), Palma de Mallorca, Balearic Islands
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - ICO Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Reina Sofía de Córdoba, Córdoba
  - Fundación Jiménez Díaz, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Virgen de la Salud de Toledo, Toledo
  - Hospital Clínico de Valencia, Valencia
  - Hospital La Fe de Valencia, Valencia

REFERENCES:
- See also: PETHEMA Foundation — http://fundacionpethema.es